CLINICAL TRIAL: NCT03328598
Title: Implementation of a Community-based Resilience Promotion Program to Only-child Loss Parents in China
Brief Title: A Community-based Resilience Program of Only-child Loss Parents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Don't have enough funding to finish the project.
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Anni Wang, Dr., Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Central South University
Record Dates: First submitted 2017-10-19; First posted 2017-11-01 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Resilience,Psychological; Bereavement; Happiness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive psychology therapy group (Experimental): This arm will be given a positive psychological group intervention developed from an foreign psychotherapy.
  Interventions: Behavioral: Positive psychology therapy group
- Resilience promotion therapy group (Experimental): This arm will be given a resilience group intervention developed from our pervious research results.
  Interventions: Behavioral: Resilience promotion therapy group
- Controlled routine activity group (Active Comparator): This arm will continue to participate in conventional community activities.
  Interventions: Other: Controlled routine activity

INTERVENTIONS:
Behavioral: Positive psychology therapy group — This program is developed from a foreign group program based on positive psychology. The positive psychology therapy lasts 8 weeks, and has a group intervention in each week. The themes of each week are start-up, time gift, positive mind, three good things, a thankful heart, life train, active service, end-up.
  Arms: Positive psychology therapy group
Behavioral: Resilience promotion therapy group — The other one is developed from research team's previous research results. The resilience promotion therapy lasts 8 weeks, and also has a group intervention in each week. The themes of each week are start-up, mutual help, trust in yourself, thanksgiving feedback, care for yourself, emotional management, end-up.
  Arms: Resilience promotion therapy group
Other: Controlled routine activity — Conventional community activities is viewed as an active comparator for controlled group.
  Arms: Controlled routine activity group

SUMMARY:
This is a community-based participatory research aiming at helping the only-child loss parents to be happier and resilient from bereavement. It is a psycho-behavioral intervention research. There are two intervention programs in this study. One is derived from a foreign psychotherapy, developed by an American psychologist and has been testified the effectiveness in promoting happiness. Another one is developed by the researchers based on the previous cross-sectional survey and interviews with those bereaved parents. The researchers will apply randomized controlled trial to testify and compare those two intervention programs in a Chinese community.

ELIGIBILITY:
Inclusion Criteria(made according to the official documents):

1. has given birth to only one child;
2. now has no living birth or adopted child;
3. the bereaved mother is older than 49 years in this family(medically maximum age for fertility in China).

Exclusion Criteria:

1. with serious mental disorders or physical illnesses;
2. are not able to complete the intervention;
3. are not able to finish questionnaire;
4. with chewing functional disorder to collect saliva dehydroepiandrosterone.

Min Age: 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Change of psychological resilience | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  Psychological resilience is a kind of ability to bounce back from adversity measured by Connor-Davidson Resilience Scale (CD-RISC).It is a self-reported scale by adding up 25 items and the total score ranges from 0-100, with higher score reflects higher resilience. The differences within two times frame are the changes of psychological resilience.

SECONDARY OUTCOMES:
Change of depression | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  Depression may refer to depressive mood in recent two weeks at each assessment measured by Zung Self-rating Depression Scale (SDS).It is a self-reported scale by adding up 20 items and the total score ranges from 20-80, with higher score reflects higher depression. The differences within time frames are changes of depression.
Change of subjective well-being | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  A feeling of happiness measured by Campbell Index of well-being (IWB).It is a self-reported scale by adding up 8 items and the total score ranges from 2.1-14.7, with higher score reflects higher subjective well-being. The differences within time frames are change of subjective well-being.
Change of social avoidance | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  The phenomenon that a person is absent from normal social interaction with others measured by Social Avoidance and Distress Scale(SAD). It is a self-reported scale by adding up 14 items and the total score ranges from 0-14, with higher score reflects social avoidance. The differences within two time frame are the changes of social avoidance.
Change of sleeping quality | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  The sleeping quality is a response of one's mood in recent month measured by Pittsburgh sleep quality index(PSQI). It is a self-reported scale, with total score higher than 19 reflects sleeping disorder. The differences within each time frames are the changes of sleeping quality.
Change of post-traumatic growth | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  The positive growth after an adversity measured by Post Traumatic Growth Inventory(PTGI). It is a self-reported scale by adding up 24 items and the total score ranges from 0-120, with higher score reflects more growth. The differences within time frames are changes of post-traumatic growth.
Change of health care behavior | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  A person's self-care behavior measured by Health Promoting Lifestyle Profile-Ⅱ( HPLP-Ⅱ).It is a self-reported scale by adding up 40 items in four dimensions. The total score ranges from 40-160, with higher score reflects better health care behavior. The differences within time frames are changes of health care behavior.
Change of concentration of dehydroepiandrosterone in saliva | Pre-intervention, post-intervention, 3 month after finishing intervention, 1 year after finishing intervention
  A kind of hormone that reflects the person's psychological stress collected by Sarstedt(Brand name) saliva collection tube by chewing the sterile cotton strips for 60 seconds. It will be tested by enzyme-linked immunosorbent assay (ELISA) with Kit Number of HT81012 and Origin site in Canada PLlabs(Company name). The differences within time frames are changes of dehydroepiandrosterone concentration in saliva.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Central South University, Changsha, Hunan
  - Yangguang Tianshi Care Center, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided
In our previous field investigation, most participants, as a vulnerable goup, are not willing to share their personal data to the public. Hence, we are not sure whether the recruited participants will agree to share the data.

REFERENCES:
- [Background] Ong AD, Bergeman CS, Bisconti TL, Wallace KA. Psychological resilience, positive emotions, and successful adaptation to stress in later life. J Pers Soc Psychol. 2006 Oct;91(4):730-49. doi: 10.1037/0022-3514.91.4.730. PMID 17014296
- [Background] Jonas-Simpson C, Steele R, Granek L, Davies B, O'Leary J. Always with me: understanding experiences of bereaved children whose baby sibling died. Death Stud. 2015 Jan-Jun;39(1-5):242-51. doi: 10.1080/07481187.2014.991954. Epub 2014 Dec 31. PMID 25551421
- [Background] Rosenberg AR, Starks H, Jones B. "I know it when I see it." The complexities of measuring resilience among parents of children with cancer. Support Care Cancer. 2014 Oct;22(10):2661-8. doi: 10.1007/s00520-014-2249-5. Epub 2014 Apr 23. PMID 24756554
- [Background] Stevens GJ, Dunsmore JC, Agho KE, Taylor MR, Jones AL, van Ritten JJ, Raphael B. Long-term health and wellbeing of people affected by the 2002 Bali bombing. Med J Aust. 2013 Mar 18;198(5):273-7. doi: 10.5694/mja12.11480. PMID 23496405
- [Background] Bonanno GA, Wortman CB, Lehman DR, Tweed RG, Haring M, Sonnega J, Carr D, Nesse RM. Resilience to loss and chronic grief: a prospective study from preloss to 18-months postloss. J Pers Soc Psychol. 2002 Nov;83(5):1150-64. doi: 10.1037//0022-3514.83.5.1150. PMID 12416919
- [Background] Sanderson C, Lobb EA, Mowll J, Butow PN, McGowan N, Price MA. Signs of post-traumatic stress disorder in caregivers following an expected death: a qualitative study. Palliat Med. 2013 Jul;27(7):625-31. doi: 10.1177/0269216313483663. Epub 2013 Apr 11. PMID 23579259
- [Background] Galatzer-Levy IR, Bonanno GA. Beyond normality in the study of bereavement: heterogeneity in depression outcomes following loss in older adults. Soc Sci Med. 2012 Jun;74(12):1987-94. doi: 10.1016/j.socscimed.2012.02.022. Epub 2012 Mar 20. PMID 22472274
- [Background] Chi P, Slatcher RB, Li X, Zhao J, Zhao G, Ren X, Zhu J, Stanton B. Perceived Stigmatization, Resilience, and Diurnal Cortisol Rhythm Among Children of Parents Living With HIV. Psychol Sci. 2015 Jun;26(6):843-52. doi: 10.1177/0956797615572904. Epub 2015 Apr 17. PMID 25888685
- [Background] Seligman MEP, Rashid T, Parks AC. Positive psychotherapy. Am Psychol. 2006 Nov;61(8):774-788. doi: 10.1037/0003-066X.61.8.774. PMID 17115810
- [Background] Seligman ME. Authentic happiness: Using the new positive psychology to realize your potential for lasting fulfillment(Simon and Schuster,2004.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/98/NCT03328598/Prot_SAP_000.pdf